CLINICAL TRIAL: NCT04610840
Title: Single-center Randomized Study to Evaluate the Safety and Effectiveness of Direct Puncture of the Caliceal System in Minipercutaneous Nephrolithotripsy (Mini-PCNL)
Brief Title: The Use of Direct Puncture Technique With Mini-PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/20-н
Record Dates: First submitted 2020-08-05; First posted 2020-11-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Urolithiasis
Keywords: urolithiasis; PCNL; direct puncture
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct puncture (Active Comparator): Direct puncture of the caliceal system performed under ultrasound or Xray control
  Interventions: Procedure: Puncture of the caliceal system
- Non-direct puncture (Active Comparator): Puncture of the caliceal system performed under ultrasound or Xray control and retrograde contrast
  Interventions: Procedure: Puncture of the caliceal system

INTERVENTIONS:
Procedure: Puncture of the caliceal system — Puncture of the caliceal system under ultrasound/Xray control

SUMMARY:
* A single-center randomized study to evaluate the safety and effectiveness of direct puncture of the caliceal system in mini-percutaneous nephrolithotripsy.
* 60 patients
* Inclusion criteria:

  1. all patients aged 18 to 70 years who are planning mini-PCNL, ready to consent to the study
  2. ASA scale 1-3
  3. Solitary stone up to 2.5 cm
  4. Single access to the caliceal system
* Exclusion criteria:

  1. Active infectious process
  2. Coagulopathies
  3. Abnormalities of the urinary system

DETAILED DESCRIPTION:
All patients will be randomized into 2 groups:

Direct puncture - patients who underwent directive puncture under ultrasound or Rg control. The number of patients is 30 people.

Non-direct puncture - patients who underwent a PCS puncture with retrograde contrast. The number of patients is 30 people.

Patients will be assigned a randomization number that matches their treatment. Block randomization using 10 blocks will be performed by a central randomization organization (www.randomize.net) using a computerized algorithm.

Primary assessed indicators:

1. Gender
2. Age
3. Body mass index
4. Localization of the stone (side, pelvis, upper anterior cup, upper posterior cup, middle anterior cup, middle posterior cup, lower anterior cup, lower posterior cup)
5. Density of the stone
6. The presence of hydronephrosis

Indicators assessed during the operation - will be assessed by the physician-researcher:

1. Installation of the ureteral catheter
2. Duration of puncture
3. Puncture method (ultrasound, X-ray)
4. The success of the insertion of a flexible guidewire into the calyceal system
5. Problems during dilation of the puncture course
6. Visualization (Excellent, Moderate, Poor)
7. Type of drainage (stent, nephrostomic tube) at the end of the operation Using the Visual Analogue Pain Scale (VAS), pain assessment is planned at 2 hours, 6 hours, 12 hours and 24 hours after surgery.

In the postoperative period, the patient independently controls the intake of analgesics from the NSAID group (ketorolac 100 mg) (Patient-controlled analgesia). If the patient requires analgesics, the time of taking the drug will be recorded (pain relief on demand).

Secondary Assessment: Postoperative Assessment

1. Complications (Clavien)
2. Hemoglobin level 24 hours after surgery
3. Creatinine level 24 hours after surgery
4. Assessment of Stone-Free status after surgery by performing multislice computed tomography of the kidneys and urinary tract without intravenous contrast

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years who are scheduled for mini-PCNL, ready to consent to the study
* ASA scale 1-3
* Solitary kidney stone up to 2.5 cm
* One access to the caliceal system

Exclusion Criteria:

* Active infectious process
* Coagulopathies
* Abnormalities of the urinary system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Puncture duration | during the operation (mini-PCNL)
  Measurement of puncture duration (in seconds)
Number of patients with successful direct puncture | during the operation (mini-PCNL)
  Evaluation of efficacy
Purity of a visual intraoperative field | during the operation (mini-PCNL)
  Excellent, Moderate, Poor visualization
Body pain | 24 hours after operation
  Using the Visual Analogue Pain Scale (VAS), pain assessment is planned at 2 hours, 6 hours, 12 hours and 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov Saint Petersburg University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No